CLINICAL TRIAL: NCT02507167
Title: Impact of Two Genetic Variants of OATP 1B3 or MRP 2 or Rifampin Mediated Transporter Inhibition on Systemic Disposition and Biological Efficacy of CCK-8 in 36 Healthy Male Individuals
Brief Title: Impact of Two Genetic Variants of OATP1B3 or MRP2 or Rifampin on Systemic Disposition and Biological Efficacy of CCK-8
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCK8/RIFA-2012
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Hormones
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mixed meal (Placebo Comparator)
  Interventions: Dietary Supplement: mixed meal
- mixed meal 2 h after single dose rifampin (600 mg) (Active Comparator)
  Interventions: Dietary Supplement: mixed meal; Drug: Rifampin

INTERVENTIONS:
Dietary Supplement: mixed meal — 250 ml Fortimel compact (chocolate)
Drug: Rifampin — oral rifampin administration (600 mg EREMFAT®)
  Arms: mixed meal 2 h after single dose rifampin (600 mg)

SUMMARY:
The purpose of this study is to evaluate the impact of genetic variants of OATP 1B3 or MRP 2 on the systemic disposition of endogenously formed CCK-8 and to determine the influence of a single-dose of the transporter inhibitor rifampin (600 mg) on the systemic disposition of endogenously formed CCK-8. Endogenous CCK-8 secretion will be induced by a single-dose standardized liquid mixed meal.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-45 years
* sex: male
* 12 subjects being homozygote wild-type carriers of OATP 1B3 (c.SLCO 1B3 699 AA and c.SLCO 1B3 334 GG) and MRP 2
* 12 subjects being homozygotes of the MRP 2 variants (genetic loss of function) and homozygote wild-type carriers of OATP 1B3
* 12 subjects being homozygotes of the OATP 1B3 variants (c.SLCO 1B3 699 GG and c.SLCO 1B3 334 TT) and homozygotes wild-type carriers of MRP 2
* BMI: ≥ 19 kg/m2 and ≤ 27 kg/m2
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which will be judged by the clinical investigator not to differ in a clinical relevant way from the healthy state
* written informed consent given by the volunteer after being provided with detailed information (both, verbally and written) about the nature, risks, and scope of the clinical trial as well as the expected desirable and adverse effects of the drug

Exclusion Criteria:

* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* gastrointestinal diseases and/or pathological findings (e.g. stenoses), which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* subjects with existing dysfunction in regulation of glucose metabolism, e.g. deficiency of glucose-6-phosphate dehydrogenase (Glc-6-P DHG) and/ or pathological findings
* subjects with alcohol and/ or drug dependence and a alcohol consumption more than 20 g alcohol/ day
* excessive smoking (more than 10 cigarettes or equivalents/ day)
* subjects with positive finding of HBsAG, HIV and/ or drugs
* subjects being on a diet (inclusive special or uniform nutritional habits, e.g. vegetarians or undercaloric diet)
* strong coffee and/ or tea consumption (≥ 1 liter a day)
* subjects suspected or known not to follow instructions
* subjects who are unable to understand written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* subjects liable to orthostatic dysregulation, fainting, or blackout
* subjects who took part in other clinical trials in the last 3 months (blocking time due to another clinical trial with investigational products)
* acute illness less than 14 d in the past
* blood donation within the last 3 months
* any medication within 4 weeks prior to the intended first administration of the study medication which might influence functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors, anticholinergics)
* any other medication within 2 weeks prior to the first administration of the study medication or less than 10-time the half-live of the respective drug
* intake of grapefruit containing food or beverages and poppy seeds containing products 14 d prior to the first drug administration until the last blood sampling of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
CCK-8 | 3 h 15 min up to 2 h 15 min before and 5, 10, 15, 20, 25, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4 h after mixed meal
  Cholecystokinin amino acid 8 concentration in blood plasma

SECONDARY OUTCOMES:
GLP-1 | 3 h 15 min up to 2 h 15 min before and 5, 10, 15, 20, 25, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4 h after mixed meal
  Glucagon-like peptide-1 concentration in blood plasma
GIP | 3 h 15 min up to 2 h 15 min before and 5, 10, 15, 20, 25, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4 h after mixed meal
  Gastric inhibitory polypeptide concentration in blood plasma
glucagon | 3 h 15 min up to 2 h 15 min before and 5, 10, 15, 20, 25, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4 h after mixed meal
  glucagon concentration in blood plasma
glucose | 3 h 15 min up to 2 h 15 min before and 15, 30, 45 min, 1, 1.25 h after mixed meal
  glucose concentration in blood plasma
potassium | 3 h 15 min up to 2 h 15 min before and 15, 30, 45 min, 1, 1.25 h after mixed meal
  potassium concentration in blood plasma
C-peptide | 3 h 15 min up to 2 h 15 min before and 15, 30, 45 min, 1, 1.25 h after mixed meal
  connecting peptide concentration in blood plasma
insulin | 3 h 15 min up to 2 h 15 min before and 15, 30, 45 min, 1, 1.25 h after mixed meal
  insulin concentration in blood plasma

OTHER OUTCOMES:
area under the curve AUC from zero to the last sampling time above the limit of quantitation (AUC0-t) of rifampin and DAc-RIF (25-O-desacetyl-rifampin) | 3 h 15 min up to 2 h 15 min, 1.5, 1 h before and 5 min, 1, 2, 3, 4, 6, 8, 10 and 14 h after mixed meal
area under the curve AUC from zero to 4 h (AUC0-4h) of rifampin and DAc-RIF (25-O-desacetyl-rifampin) | 3 h 15 min up to 2 h 15 min, 1.5, 1 h before and 5 min, 1, 2 h after mixed meal
maximal concentration (Cmax) of rifampin and DAc-RIF (25-O-desacetyl-rifampin) | 3 h 15 min up to 2 h 15 min, 1.5, 1 h before and 5 min, 1, 2, 3, 4, 6, 8, 10 and 14 h after mixed meal
time point of maximal concentration (tmax) of rifampin and DAc-RIF (25-O-desacetyl-rifampin) | 3 h 15 min up to 2 h 15 min, 1.5, 1 h before and 5 min, 1, 2, 3, 4, 6, 8, 10 and 14 h after mixed meal
terminal half-life (t1/2) of rifampin and DAc-RIF (25-O-desacetyl-rifampin) | 3 h 15 min up to 2 h 15 min, 1.5, 1 h before and 5 min, 1, 2, 3, 4, 6, 8, 10 and 14 h after mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Greifswald, Germany